CLINICAL TRIAL: NCT02771288
Title: Safety and Vascular Remodelling After Bioresorbable Vascular Scaffold Implantation for Stenotic or Occluded Lesions in Children and Young Adults With Kawasaki Disease
Brief Title: Safety and Vascular Remodelling After BVS Implantation for Stenotic or Occluded Lesions in Children and Young Adults With KD.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201512126DINC
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Kawasaki Disease
Keywords: Kawasaki disease; optical coherence tomography; multislice computed tomography
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kawasaki disease (Other)
  Interventions: Device: Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Bioresorbable Vascular Scaffold

SUMMARY:
To investigate the safety and long-term vascular remodeling after bioresorbable vascular scaffold (BVS) implantation for stenotic or occluded lesion in children or young adults with Kawasaki disease (KD).

Background: KD occurs worldwide, most prevalent in Japan and East Asian countries. Coronary artery lesion is the predominant determinant of KD outcome in the long-term. Children with KD with aneurysms at least 6 mm in maximal diameter had a greater than 50% chance of developing a clinically significant stenotic lesion during follow-up. They are at risk of myocardial infarction-related sudden death or congestive heart failure as young adults. Bypass surgery could be the reasonable strategy but the long-term patency of the graft remains unsatisfactory. Percutaneous angioplasty with drug-eluting stents (DES) implantation is the alternative. However, metallic stenting remains problematic in several aspects mainly due to the restriction of vessel expansive remodeling. The novel BVS has the potential to be free from the limitation due to scaffold degradation.

DETAILED DESCRIPTION:
we will conduct a single-center, single-group prospective study with safety and imaging endpoints. A total of 10 KD children or young adults with indication of revascularization are enrolled, and BVS will be implanted for stenotic or occluded lesions. QCA and optical coherence tomography (OCT) are used to evaluate the baseline lumen area, plaque characteristics, and BVS expansion or eccentricity after deployment. At 12 months, scaffold restenosis is evaluated by multislice computed tomography. At 30 months, patients will receive follow-up by angiography and OCT to evaluate lumen area, neoplaque characteristics, and side branch conditions. Otherwise, the composite endpoint including cardiac death, myocardial infarction, and ischaemia-driven target lesion revascularisation are assessed at 30 days, 6 and 9 months, and 1, 2, 3 years.

ELIGIBILITY:
Inclusion criteria:

1. In the single-group prospective study with safety and imaging endpoints, a total of 10 KD patients < 18 years will be enrolled.
2. The diagnosis of KD was made based on clinical criteria for KD.

Exclusion criteria:

Patients presenting with an acute myocardial infarction or unstable arrhythmias, or those who has severe left ventricular dysfunction (ejection fraction less than 35%), intrastent restenotic lesions, lesions located in the left main coronary artery, and tight lesions which could not be well dilated even after rotational atherectomy are excluded. Those with chronic renal insufficiency (creatinine >1.5 mg/dl) are also excluded due to the limitation of OCT (optical coherence tomography) use.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
time to disease progression | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yi-Chih, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan

IPD SHARING:
Plan to Share IPD: No